CLINICAL TRIAL: NCT03508830
Title: Minimally Invasive Thoracic Surgery Intercostal Nerve Block Trial - Liposomal Bupivacaine Versus Standard Bupivacaine
Brief Title: Minimally Invasive Thoracic Surgery Intercostal Nerve Block Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Johannes R. Kratz, MD, Assistant Professor of Surgery Division of Adult Cardiothoracic Surgery; Van Auken Endowed Chair in Thoracic Oncology; Director, Minimally Invasive and Robotic Thoracic Surgery; Associate Director, Thoracic Surgery Residency Program, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P0530291
Record Dates: First submitted 2018-03-23; First posted 2018-04-26 (Actual); Results first posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Thoracic Diseases; Postoperative Pain; Opioid Use
Keywords: Liposomal Bupivacaine; Intercostal Nerve Block; Minimally Invasive Thoracic Surgery
MeSH Terms: conditions — Thoracic Diseases; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Syringe with Obscuring Over-Wrap
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liposomal Bupivacaine (Experimental): 5cc of drug preparation will be percutaneously injected into each intercostal space 3-10 under direct intrathoracic vision and subcutaneously into each surgical wound at the conclusion of the surgery.
  Drug Preparation: 266mg (20cc) Liposomal Bupivacaine admixed with 0.25% (2.5mg/cc) Standard Bupivacaine (maximum dose of 2mg/kg) and varied 0.9% normal saline volume for total volume of 60cc.
  Interventions: Drug: Liposomal bupivacaine
- Standard Bupivacaine (Active Comparator): 5cc of drug preparation will be percutaneously injected into each intercostal space 3-10 under direct intrathoracic vision and subcutaneously into each surgical wound at the conclusion of the surgery.
  Drug Preparation - 0.25% (2.5mg/cc) Standard Bupivacaine (maximum dose of 2mg/kg) admixed with varied 0.9% normal saline volume for total volume of 60cc.
  Interventions: Drug: Bupivacaine Injection

INTERVENTIONS:
Drug: Liposomal bupivacaine — 5cc of drug preparation will be percutaneously injected into each intercostal space 3-10 under direct intrathoracic vision and subcutaneously into each surgical wound at the conclusion of the surgery.
  Arms: Liposomal Bupivacaine
Drug: Bupivacaine Injection — 5cc of drug preparation will be percutaneously injected into each intercostal space 3-10 under direct intrathoracic vision and subcutaneously into each surgical wound at the conclusion of the surgery.
  Arms: Standard Bupivacaine

SUMMARY:
The Minimally Invasive Thoracic Surgery Intercostal Nerve Block Trial is a single center, double-blind, randomized, active-comparator controlled clinical trial to assess the analgesic efficacy of intercostal nerve block by Liposomal Bupivacaine versus Standard Bupivacaine in subjects undergoing lung resection by robotic or video-assisted thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Robotic or Video-Assisted Lung Resection for All Indications

Exclusion Criteria:

* Additional Thoracic Procedures (beyond lung resection and mediastinal lymphadenectomy)
* Extra-Thoracic Procedures
* Hypersensitivity to Amide Local Analgesia
* Cardiac Conduction Abnormalities
* Hepatic Dysfunction
* Preoperative Neuropathic Pain and/or Preoperative Daily Opioid Usage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-12-30 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Liposomal Bupivacaine: Liposomal Bupivacaine: Drug percutaneously injected into intercostal spaces 3-10 under direct intrathoracic vision.
- Standard Bupivacaine: Standard Bupivacaine: Drug percutaneously injected into intercostal spaces 3-10 under direct intrathoracic vision.
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Started | 46 | 45
Completed | 41 | 39
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Physician Decision | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [62 to 77] | 67 [62 to 77] | 69 [62 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 12 | 10 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 29 | 28 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 39 | 80
Smoker [Count of Participants; unit: Participants] | 21 | 23 | 44
Primary Lung Cancer [Count of Participants; unit: Participants] | 35 | 36 | 71
Robotic Surgery [Count of Participants; unit: Participants] | 39 | 39 | 78
Sublobar Resection [Count of Participants; unit: Participants] | 32 | 28 | 60

OUTCOME MEASURES:

1. Primary Outcome: Average Daily In-Hospital Use of Opioids
Description: Measured in Oral Morphine Equivalents per Day
Time Frame: Average over Entire Length of Hospitalization (Up to 1 Week)
Measure: Mean (Standard Deviation); unit: Oral Morphine Equivalent per Day
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 41 | 39
Oral Morphine Equivalent per Day | 40 (28) | 45 (27)

2. Secondary Outcome: Average Daily In-Hospital Pain Score
Description: Measured 0-10 Visual Analog Scale for Pain (Higher Score Means Worse Pain).
Time Frame: Average over Length of Hospitalization - Up to 1 Week
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 41 | 39
Units on a Scale | 2.7 (1.7) | 3.1 (1.7)

3. Secondary Outcome: Number of Participants With Postoperative Pneumonia
Description: Pneumonia (Y/N)
Time Frame: Index Hospitalization following Surgery until Discharge - Up to 1 Week
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 41 | 39
Participants | 0 | 1

4. Secondary Outcome: Length of Stay
Description: Measured in Days
Time Frame: Index Hospitalization following Surgery until Discharge - Up to 1 Week
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 41 | 39
Days | 2.2 (1.1) | 2.3 (1.3)

ADVERSE EVENTS:
Time Frame: From time of drug administration to subsequent 30 days.
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/39
Other Adverse Events (participants affected / at risk) | 0/41 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT03508830/Prot_SAP_000.pdf